CLINICAL TRIAL: NCT01172964
Title: A Pilot Feasibility Study of Oral 5-Fluorocytosine and Genetically-Modified Neural Stem Cells Expressing E.Coli Cytosine Deaminase for Treatment of Recurrent High Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08002; NCI-2010-01388 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Adult Anaplastic Astrocytoma; Recurrent Grade III Glioma; Recurrent Grade IV Glioma; Adult Anaplastic Oligodendroglioma; Adult Brain Tumor; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Recurrent Adult Brain Tumor; Adult Anaplastic Oligoastrocytoma; Recurrent High Grade Glioma
Keywords: Los Angeles
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Brain Neoplasms; Glioblastoma; Gliosarcoma; Glioma | interventions — Flucytosine; Polymerase Chain Reaction; Immunohistochemistry; Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo debulking craniotomy and receive injections of HB1.F3.CD neural stem cells directly into brain tissue on day 0. Patients then receive oral 5-fluorocytosine every 6 hours on days 4-10 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: flucytosine; Other: polymerase chain reaction; Other: immunohistochemistry staining method; Biological: gene therapy; Other: pharmacological study; Other: 3-Tesla magnetic resonance imaging; Other: laboratory biomarker analysis; Procedure: therapeutic conventional surgery; Biological: E. coli CD-expressing genetically modified neural stem cells

INTERVENTIONS:
Drug: flucytosine — Given orally
  Other Names: 5-FC; 5-fluorocytosine; Alcobon; Ancobon; Ancotil; Ro 2-9915
Other: polymerase chain reaction — Correlative studies
  Other Names: PCR
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Biological: gene therapy — Injected at the time of the surgery to resect the tumor
  Other Names: therapy, gene
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: 3-Tesla magnetic resonance imaging — Correlative studies
  Other Names: 3-Tesla MRI; 3T MRI
Other: laboratory biomarker analysis — Correlative studies
Procedure: therapeutic conventional surgery — Surgery to resect the tumor
Biological: E. coli CD-expressing genetically modified neural stem cells — Injected at the time of the surgery to resect the tumor
  Other Names: HB1.F3.CD neural stem cells

SUMMARY:
RATIONALE: Genetically-modified neural stem cells (NSCs) that convert 5-fluorocytosine (5-FC) into the chemotherapy agent 5-FU (fluorouracil) at sites of tumor in the brain may be an effective treatment for glioma.

PURPOSE: This clinical trial studies genetically-modified NSCs and 5-FC in patients undergoing surgery for recurrent high-grade gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of intracerebral administration of NSCs in combination with oral 5-FC in patients with recurrent high-grade gliomas.

SECONDARY OBJECTIVES:

I. To characterize the relationship between intracerebral and systemic concentrations of 5-FC and 5-FU with increasing NSC dose level.

II. To non-invasively assess the presence of 5-FU in the brain with the use of fluorine (19F)-magnetic resonance spectroscopy (MRS)(no longer in effect as of 5/1/2012).

III. To assess for the possible development of immunogenicity against the NSCs.

IV. To assess the intracerebral distribution of NSCs using iron-labeling as a cellular tracker.

V. To gather preliminary imaging data regarding perfusion permeability parameters and imaging characteristics as shown on magnetic resonance imaging (MRI) studies due to the presence of NSCs in the brain.

VI. To determine, at time of autopsy, the fate of the NSCs.

OUTLINE:

This is a dose-escalation study.

After biopsy or surgery to resect tumor, study patients receive injections of genetically modified NSCs directly into brain tissue on day 0. Patients then take oral 5-FC every 6 hours during days 4-10 which is converted to 5-FU in the brain by the NSCs.

Follow-up MRIs of the brain are performed on days 32, 60, and every 2 months thereafter to assess for response and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient has had a prior, histologically-confirmed, diagnosis of a grade III or grade IV glioma (including glioblastoma, anaplastic astrocytoma, gliosarcoma, anaplastic oligodendroglioma, or anaplastic oligoastrocytoma), or has a prior, histologically-confirmed, diagnosis of a grade II glioma and now has radiographic findings consistent with a high-grade glioma (grade III or IV)
* Imaging studies show evidence of recurrent supratentorial tumor(s)
* The patient must be in need of a craniotomy for tumor resection or a stereotactic brain biopsy for the purpose of diagnosis or differentiating between tumor progression versus treatment-induced effects following radiation therapy +/- chemotherapy
* Based on the neurosurgeon's judgment, there is no anticipated physical connection between the post-resection tumor cavity and the cerebral ventricles
* Patient's high-grade glioma has recurred or progressed after chemoradiation
* Patient has a Karnofsky Performance Status of >= 70%
* Patient has a life expectancy of >=3 months
* If patient requires corticosteroids for the control of cerebral edema, s/he must be on a stable dose for at least 1 week prior to enrollment
* Patient has recovered from toxicity of prior therapies; an interval of at least 12 weeks must have elapsed since the completion of radiation therapy; at least 6 weeks since the completion of nitrosourea-containing chemotherapy regimen; and at least 4 weeks since the completion of a non-nitrosourea-containing cytotoxic chemotherapy regimen; if a patient's most recent treatment was with a targeted agent only; and s/he has recovered from any toxicity of this targeted agent, then a waiting period of only 2 weeks is needed from the last dose and the start of study treatment, with the exception of bevacizumab where a wash out period of at least 4 weeks is required before starting study treatment
* Absolute neutrophil count of >= 1,500 cells/mm^3 and platelet count >= 100,000 cells/mm^3
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 4 times the institutional upper limit of normal
* Serum creatinine =< the institutional upper limit of normal
* Patients must be able to swallow pills
* Patients must be able to understand and be willing to sign a written informed consent document
* Female patients of child-bearing potential and sexually active male patients must agree to use an effective method of contraception while participating in this study
* Women of childbearing potential must have a negative pregnancy =< 2 weeks prior to registration

INCLUSION CRITERIA FOR PROCEEDING TO TREATMENT WITH 5-FC:

* Patients must be tolerating oral intake
* Patients' daily total dose of dexamethasone must be < 12 mg by Day 4

Exclusion Criteria:

* Patients who are currently receiving chemotherapy, radiotherapy, or are enrolled in another treatment clinical trial
* Patients who have anti-human leukocyte antigen (HLA) antibodies specific for HLA antigens expressed by the HB1.F3.CD NSCs
* Patients who are unable to undergo an MRI
* Patients with chronic or active viral infections of the central nervous system (CNS)
* Patients who are allergic to 5-FC or 5-FU
* Patients who have a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Female patients who are pregnant or breast-feeding
* Patients who have not recovered from the toxicities of prior chemotherapy or radiotherapy
* Patients who require anti-seizure medication but are not on a stable dose of anti-seizure medication for at least 1 week prior to enrollment

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2015-02-11 (Actual); Study Completion 2015-02-11 (Actual)

PRIMARY OUTCOMES:
Determination of the safety and feasibility of intracerebral administration of genetically-modified neural stem cells (NSCs) in combination with oral 5-fluorocytosine. | Day 60
  Measures of feasibility include the incidence of clinically symptomatic intratumoral hemorrhage, CNS infection, seizures, altered mental status, development of focal neurologic deficits, as well as chemotherapy-associated toxicities. All toxicities at each dose level will be summarized using descriptive statistics. Graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Relationship between intracerebral and systemic concentrations of 5-FC and 5-FU with increasing NSC dose level | Up to Day 10
  Summarized by NSC dose cohort using descriptive statistics and graphs. The Macdonald Criteria will be used to assess response. As of 11/30/2012 patients will no longer undergo these tests.
Presence of 5-FU in the brain using 19F-MRS | Day 60
  As of 5/1/2012, study patients will no longer undergo 19F-MRS.
Assessment of development of immunogenicity against NSCs | Day 60
  As of 11/30/2012 patients will no longer undergo these tests.
Obtain preliminary imaging data regarding perfusion permeability parameters and imaging characteristics as shown on magnetic resonance imaging (MRI) studies due to the presence of NSCs in the brain. | Day 60
Assessment of the fate of NSCs at autopsy when feasible | At autopsy
Assess the intracerebral distribution of NSCs using iron-labeling as a cellular tracker. | Up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States